CLINICAL TRIAL: NCT05068583
Title: Liquid Biopsies in Non-CNS Malignant Pediatric Solid Tumors
Brief Title: Liquid Biopsies in Pediatric Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Fariba Navid, Principle Investigator, Children's Hospital Los Angeles
Other Study IDs: CHLA-19-00146
Record Dates: First submitted 2021-08-30; First posted 2021-10-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Solid Tumor, Unspecified, Protocol Specific
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Osteosarcoma
  Interventions: Other: Blood Draw
- Ewing Sarcoma
  Interventions: Other: Blood Draw
- Rhabdomyosarcoma
  Interventions: Other: Blood Draw
- Synovial Sarcoma
  Interventions: Other: Blood Draw
- Non-Rhabdomyosarcoma Soft Tissue Sarcoma
  Interventions: Other: Blood Draw
- Hepatic Tumors
  Interventions: Other: Blood Draw
- Renal Tumors
  Interventions: Other: Blood Draw
- Thyroid Tumors
  Interventions: Other: Blood Draw
- Germ Cell Tumors
  Interventions: Other: Blood Draw
- Healthy Volunteers
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood draw at baseline, disease evaluation time point, and pre and post surgery and/or radiation.

SUMMARY:
This study is being done to determine if traces of tumor can be found in the blood before, during, and after patients stop treatment. We will analyze the tumor material to see if it is similar to tumor tissue and if the tumor material in blood is helpful in monitoring the disease.

DETAILED DESCRIPTION:
Liquid biopsies, particularly those involving cell-free DNA (cfDNA), are a promising non-invasive, cost effective method of monitoring disease in cancer patients with solid tumors and are being increasingly employed in various adult malignancies to diagnose disease, monitor tumor response, detect relapse and learn more about tumor biology. The utility of liquid biopsies which may include isolation and analysis of tumor derived material such as DNA, RNA, intact cells, proteins, or exosomes from blood or other bodily fluids in pediatric solid tumors has not been established. In this study, we propose to prospectively collect serial blood samples at baseline, during therapy, end of therapy, relapse, and during follow up from patients ≥ 6 months of age with newly diagnosed or relapsed/refractory various pediatric non-CNS malignant solid tumors to determine the feasibility of detecting various tumor-derived material, including exosomes, circulating tumor cells, and circulating tumor nucleic acid (ctDNA and ctRNA). The timing of blood sample collection will be during a routine lab draw around the time of a disease evaluation. The ctDNA and ctRNA as well as DNA and RNA extracted from tumor-derived exosomes will be quantified at each time point and the findings will be correlated with conventional methods for disease evaluation (e.g., imaging studies, histologic tumor response, or serum tumor markers) and outcome (overall survival and event-free survival).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, relapsed, or refractory histologically confirmed high grade bone or soft tissue sarcoma or malignant renal, thyroid, germ cell, or hepatic tumors, OR
* Healthy individual with no history of cancer or chronic medical problems and < 21 years of age

Exclusion Criteria:

* CNS Malignancies
* Individuals < 6 months of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients over the age of 6 months who are newly diagnosed, relapsed, or refractory histologically confirmed high grade bone or soft tissue sarcoma or malignant renal, thyroid, germ cell, or hepatic tumors. Also, healthy individuals with no history of cancer or chronic medical problems who are < 21 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2029-05-08 (Estimated); Study Completion 2034-05-08 (Estimated)

PRIMARY OUTCOMES:
To detect circulating tumor DNA (ctDNA) in serial blood samples from patients with pediatric non-CNS solid tumors using low pass whole genome sequencing. | 10 years
  To determine how often circulating tumor DNA (ctDNA), circulating tumor cells (CTCs), and circulating tumor RNA (ctRNA) is detected in serial blood samples from patients with newly diagnosed and relapsed/refractory malignant pediatric solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Navid, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
For patients that are alive, we do not plan to share IPD.